CLINICAL TRIAL: NCT04150406
Title: Flexofytol®, a Curcuma Extract, for the Treatment of Endometriosis- Associated Pain: a Randomized, Double Blind, Placebo-controlled Study
Brief Title: Flexofytol® for the Treatment of Endometriosis- Associated Pain
Acronym: ENDOFLEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Alexandra Perricos, Principal investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1712/2019
Record Dates: First submitted 2019-10-29; First posted 2019-11-04 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Endometriosis
Keywords: Curcuma; Endometriosis-associated pain
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexofytol (Active Comparator): 2 capsules containing 42mg of curcumin will be administered twice a day for a duration of 4 months.
  Interventions: Dietary Supplement: Flexofytol
- Placebo (Placebo Comparator): 2 capsules of the placebo, identical in appearance to Flexofytol, will be administeres twice a day for a duration of 4 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Flexofytol — Curcuma extract
  Arms: Flexofytol
Other: Placebo — placebo
  Arms: Placebo

SUMMARY:
Endometriosis is a benign disease that affects 6-10% of women of reproductive age. The wide range of symptoms observed in patients with endometriosis is due to implantation of endometrial tissue outside the uterine cavity. This ectopic endometrium is subjected to cyclic changes similar to that of eutopic endometrium. Typically, ectopic lesions are found in the pelvis, notably on the ovaries in the form of cysts (endometriomas), as well as the rectouterine and vesicouterine pouch. Lesions have also been described in other parts of the abdomen and in other locations outside the abdominal cavity.

Although endometriosis has also been described in asymptomatic patients, possible symptoms range from mild to severe pain presenting itself as dysmenorrhea, dyspareunia, or dyschezia, or as infertility. Since the clinical picture varies, the treatment of this disease has become quite personalized. Many studies conducted over the past several years have presented different treatment options for the symptoms caused by endometriosis.

Turmeric, which is won from the rootstalks of Curcuma longa, has more than 300 biologically active elements. One of the three main curcuminoids that are derived from turmeric, is curcumin. Several in-vitro and animal studies have described anti-oxidant, anti-inflammatory and anti-angiogenic effects of curcumin.

The main objective for the treatment of endometriosis patients is symptom relief. Treatment options include analgesic therapies, hormonal therapies, laparoscopic surgery or a combination of these. For patients who refuse hormonal therapies however, conservative treatment options are limited.

Curcuma is a substance that has been in use for centuries, especially in ayurvedic and Traditional Chinese Medicine for the treatment of various symptoms, notably for pain alleviation in inflammatory illnesses. Several recently published studies have shown very promising results of Flexofytol for pain alleviation in patients with osteoarthritis, due to its anti-inflammatory and anti-oxidant properties. Due to these properties of curcuma, we aim to analyse if curcuma capsules, sold by the pharmaceutical company Tilman under the name Flexofytol®, can be used to alleviate symptoms in patients suffering from endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women between the ages of 18 and 51 years
* Ability to comprehend the full nature and purpose of the study
* Signed informed consent
* Diagnosed endometriosis (peritoneal, ovarian or deep-infiltrating endometriosis (DIE))
* By laparoscopy or laparotomy with histological verification diagnosed up to 10 years before screening
* By ultrasound or MRI (ovarian or deep-infiltrating endometriosis, as peritoneal lesions can only be evaluated surgically)
* Moderate to severe pelvic pain (i.e. dysmenorrhea or NMPP of at least 4 on the 1-10 NRS) at least during the past 3 months
* Refusal of hormonal treatments
* The patient must agree to switch from her usual analgesic rescue medication to only the one permitted by the study during screening, treatment and follow-up period

Exclusion Criteria:

* The patient is pregnant or breast feeding or is planning a pregnancy within the treatment period
* Known addiction (alcohol, drugs, pills, etc...)
* Liver or kidney problems
* Known problems of the bile system
* Infection (HIV, Hepatitis, TBC, etc..) or systemic autoimmune diseases
* Known or suspected malignant disease
* Intake of blood-thinning medication (such as heparin or aspirin for example)
* Intake of hormonal contraceptives (oral during the last 4 weeks, injectable: during the last 3 months)
* Patient with a surgical history of hysterectomy, bilateral adnexectomy, endometrial ablation resulting in amenorrhea

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of the average pain score from baseline to 4 months after begin of treatment | 4 months
  Pain will be evaluated using the Numeric Rating Scale (NRS), from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Change in number of days with pain ≥ NRS 4 from baseline to 4 months after begin of treatment | 4 months
  Pain will be evaluated using the Numeric Rating Scale (NRS), from 0 (no pain) to 10 (worst pain imaginable).
Alleviation of dyspareunia using the NRS between 0 and 10, from baseline to 4 months after begin of treatment points) | 4 months
  Pain will be evaluated using the Numeric Rating Scale (NRS), from 0 (no pain) to 10 (worst pain imaginable).
Alleviation of dysuria using the NRS between 0 and 10 points, from baseline to 4 months after begin of treatment | 4 months
  Pain will be evaluated using the Numeric Rating Scale (NRS), from 0 (no pain) to 10 (worst pain imaginable).
Alleviation of dyschezia using the NRS between 0 and 10 points from baseline to 4 months after begin of treatment | 4 months
  Pain will be evaluated using the Numeric Rating Scale (NRS), from 0 (no pain) to 10 (worst pain imaginable).
Change in quality of life (using the numerical score of the Endometriosis health profile - EHP 30) | 4 months
  evaluated using a scale of 0 - 100, where 0 indicates the best health status and 100 the worst health status
Change in sexual function (using the numerical score of the female sexual function index - FSFI) | 4 months
  each question answered using a score from 0 to 5, 0 indicating no sexual activity, and, depending on the question, 1 indicating high satisfaction or high frequency, to 5 indicating low satisfaction or low frequency.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Vienna, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No